CLINICAL TRIAL: NCT07118553
Title: The Effect of Facial Massage on Quality of Life, Mood, Pain and Stress Levels in Women With Premenstrual Syndrome
Brief Title: Factors Affecting Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trabzon University (Other)
Responsible Party: Principal Investigator, Aysun YAĞCİ ŞENTÜRK, Assistant professor, Trabzon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU-TMYO-AYŞ-01
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome; face; massage; quality of life
MeSH Terms: conditions — Premenstrual Syndrome; Facies

STUDY DESIGN:
Intervention Model Description: two groups (intervention and control groups)
Who Masked: Participant
Masking Description: The intervention group received facial massage. The control group continued their lives in the same manner. At the end of six weeks, the researchers completed post-tests for both groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial massage group (Experimental): Classical facial massage was applied to the intervention group 2 days a week (with at least 1 day break) for 6 weeks. A session continued 20-30 minutes.
  Interventions: Other: classic facial massage
- control group (No Intervention): The control group received no intervention. Participants continued their daily routines as usual.

INTERVENTIONS:
Other: classic facial massage — Powder was used as an intermediate product in facial massage application. Before the application, the participants were made to lie in the supine position on the patient's bed. The researchers performed the facial massage by standing at the participants' bedside. During the massage application, three stroking movements were applied to the chin, mouth, nose, eyes and forehead areas, respectively. Kneading motion was then applied to the same areas three times each. Then, stroking was applied to these five areas again and the facial massage application was terminated at the end of approximately 20-30 minutes. Friction movement was applied to the temporal region in each stroking and kneading application
  Arms: Facial massage group

SUMMARY:
Premenstrual pain syndrome is a common problem that affects many women of reproductive age. In this study, we aimed to determine whether facial massage would improve the quality of life, mood, pain and stress levels of women with premenstrual syndrome.

DETAILED DESCRIPTION:
Young women over the age of 18 with premenstrual syndrome were randomly divided into two groups. One group received facial massage for six weeks, while the other group received no intervention. At the end of six weeks, pain, stress, quality of life and mood were assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* at least 111 points or more on the Premenstrual Syndrome Scale
* 8 years of age or older
* to be volunteer for the study

Exclusion Criteria:

* presence of any open wounds, allergies, etc. that would prevent facial massage
* the presence of routinely used gynaecological medication
* regular exercise
* unwillingness to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | six weeks
  The VAS was used to assess participants' pain intensity. The VAS is a scale ranging from 0 ('No pain') to 10 points ('Unbearable pain') on a horizontal line. According to the VAS, '0' means no pain, while 10 points means severe pain.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | six weeks
  PSS 5-point Likert-type scale ranging from 'Never (0)' to 'Very often (4)'
  * PSS-10 takes a value between 0 and 40 points and a high score indicates a high level of stress PSS 5-point Likert-type scale ranging from 'Never (0)' to 'Very often (4)'
  * PSS-10 takes a value between 0 and 40 points and a high score indicates a high level of stress 5-point Likert-type scale ranging from 'Never (0)' to 'Very often (4)'
  * PSS-10 takes a value between 0 and 40 points and a high score indicates a high level of stress PSS is a 5-point Likert-type scale ranging from 'Never (0)' to 'Very often (4). Minimum score of the scale is 0 while the maximum score is 40. High scores indicates a high level of stress.
Short Form-12 | six weeks
  It is a short version of the Short Form-36 scale and it evaluates quality of life. An increase in the obtained score indicates a good quality of life.
Profile of Mood States (POMS): | six weeks
  POMS is a 5-point Likert scale and the response to each item is scored as never (0 points), very little (1 point), moderately (2 points), quite a lot (3 points), extremely (4 points). The total scale score is obtained by subtracting the score of the vigour-activity subscale from the total score of the other items. A high score indicates the presence of a mood disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Yağci Şentürk, Ph.D, Principal Investigator — Trabzon University
Locations (1):
- Trabzon Unversity, Trabzon, Tonya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No